CLINICAL TRIAL: NCT00284167
Title: Efficacy of a Web-based Tailored Weight Management Program With and Without Tailored Nutrition and Goal Setting Support
Brief Title: Efficacy of a Web-based Tailored Weight Management Program
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Collaborators: Kaiser Permanente (Other)
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: 49147
Record Dates: First submitted 2006-01-24; First posted 2006-01-31 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Obesity
Keywords: tailored; web-based; weight management; obesity; efficacy
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: tailored web-based weight management intervention

SUMMARY:
The primary objective of this study is to assess the benefit of using online, tailored behavioral weight management materials (Balance), in combination with nutritional materials (Balance and Nourish), in conjunction with a goal setting tool (Balance and Achieve), or a combination of all three (Balance, Nourish and Achieve). This objective will be evaluated by measuring weight loss rates as reported by study participants at 3, 12, and 18 months post-enrollment. The hypothesis is that adding additional materials will increase the effect of the intervention over just using Balance alone.

DETAILED DESCRIPTION:
This will be a randomized control, web-based trial for weight management with four treatment arms. Participants will be assigned to receive tailored materials from either: 1) the Balance program, 2) the Balance and Nourish programs, 3) the Balance and Achieve programs, or 4) the Balance, Nourish and Achieve programs. Participants will be recruited directly through their health care organization. In order to participate, participants must visit the website to confirm their eligibility, e.g. valid e-mail address. Those who wish to participate will provide consent on the Web, and then will be presented with an online questionnaire. These questions will provide baseline data for each participant and will be the basis for the tailoring of the Balance materials each participant will receive. Within 24 hours of submitting the completed questionnaire, participants will be informed by e-mail that their tailored Balance plan is available on the website. They will receive follow-up materials by e-mail during the six-week period after they enroll. Participants who have been assigned to additional programs will be sent e-mails with links to the relevant programs. At 3, 12 and 18 months, all participants will be assessed via an online survey. The assessment will include weight management parameters, psychosocial outcomes, and program utilization. This data will be self-reported.

STUDY POPULATION The study sample will be drawn from members of three integrated delivery systems: Kaiser Permanente Colorado (KPCO), Kaiser Permanente Ohio (KPOH), and Group Health Cooperative (GHC) of Puget Sound. In order to participate, participants must access and enroll in the study on the Web. A total of 1,848 participants will be enrolled within a six-month period, with approximately 450 participants in each treatment arm. By 18-month follow-up, we assume successful data collection from at least 65 percent of the enrollees, or 1200 participants, 300 in each treatment group. The study is open to those who meet the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age
2. Current KP or GHC member
3. BMI greater than or equal to 30 or BMI greater than or equal to 25 and have one of the following chronic illnesses: diabetes, coronary artery disease, depression, or asthma, or arthritis.
4. Agree to be contacted via computerized questionnaire at 3, 12 and 18 months post-enrollment
5. Regular access to the Internet and a functioning e-mail address

Exclusion Criteria:

1. Current use of pharmacologic, behavioral or surgical treatment for weight loss
2. Currently pregnant or planning pregnancy
3. Inability to read English.
4. Presence of Congestive Heart Failure
5. KP Ohio region members who participated in the original THeME study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1848
Dates: Start 2003-09; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess weight reduction at 3, 12, and 18 months post intervention.

SECONDARY OUTCOMES:
• To assess psychosocial outcomes including motivation and self-efficacy.
• To assess the degree to which participants perceive their support materials have been tailored for them.
• To assess lifestyle changes including physical activity and nutrition
• To examine relative effectiveness of web-based programs given age, gender, preferred language, ethnicity, and utilization patterns.
• To examine percent of weight loss goal attainment.
• To examine participation rates by the BMI strata stated above.
• To assess the perceived helpfulness of the behavioral support materials with the participants' weight loss attempts.
• To assess the overall satisfaction with the programs.
• To assess participant satisfaction with Kaiser Permanente or GHC.
• To assess changes in self-reported health status.
• To assess changes in self-reported medical outpatient utilization.
• To assess self-reported work productivity (days missed from work or school).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Wildenhaus, Ph.D., Principal Investigator — HealthMedia, Inc.; Russ Glasgow, Ph.D., Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Care Management Institute, Walnut Creek, California, United States